CLINICAL TRIAL: NCT05371340
Title: The Efficacy of Quercetin Supplementation on Bone Turnover Markers, Inflammatory Markers, Body Composition, and Physical Function in Post-Menopausal Women
Brief Title: Quercetin's Effect on Bone Health and Inflammatory Markers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kennesaw State University (Other)
Responsible Party: Principal Investigator, Trisha VanDusseldorp, Director, Kennesaw State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 19-476
Record Dates: First submitted 2022-05-03; First posted 2022-05-12 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Osteoporosis, Postmenopausal
Keywords: Bone turnover markers; Quercetin
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Quercetin

STUDY DESIGN:
Intervention Model Description: Double blind placebo controlled
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Postmenopausal women: Experimental group (Experimental): Quercetin 500 mg. One capsule once a day.
  Interventions: Dietary Supplement: Quercetin (500 mg)
- Postmenopausal women: Placebo group (Placebo Comparator): Placebo (methylcellulose E4M) 500 mg, once capsule once a day.
  Interventions: Other: Placebo (500 mg)

INTERVENTIONS:
Dietary Supplement: Quercetin (500 mg) — Once-daily 500 mg Quercetin
  Arms: Postmenopausal women: Experimental group
Other: Placebo (500 mg) — Once-daily 500 mg methylcellulose 9E4M)
  Arms: Postmenopausal women: Placebo group

SUMMARY:
Quercetin is a plant-based flavonoid that is naturally found in many fruits and vegetables, and is considered to be a potent antioxidant with several expected health benefits such as anti-inflammatory effects and bone-conserving properties. Participants will supplement with either Quercetin, or placebo, for 90-days with pre- and post-testing visits.

DETAILED DESCRIPTION:
Quercetin is a plant-based flavonoid that is naturally found in many fruits and vegetables such as onions, apples, berries, green tea, and red wine and is currently an FDA approved supplement. Quercetin is considered to be a potent antioxidant with several expected health benefits. Both in vivo and in vitro studies have demonstrated that quercetin acts as a potent natural osteogenic agent with benefits that include anti-inflammatory effects and bone-conserving properties. Quercetin is suggested to protect against bone loss by inhibiting bone resorption and stimulating bone formation which is indicated by an increase in bone mineral density and bone formation markers such as osteocalcin.

The purpose of this study is to investigate the effects of quercetin supplementation on bone, specifically on bone turnover markers, in postmenopausal women. The interplay between cytokines (i.e., IL-6, CRP, and TNF-alpha) and bone turnover markers was also considered.

In a double-blind, placebo-controlled fashion, we aimed to recruit 50, healthy, postmenopausal women between the ages of 45-75 years to participate in a 90-day supplement trial. Participants will be randomly assigned to one of two supplement groups: 1) quercetin 500 mg, once per day, or 2) placebo (methyl cellulose E4M) 500 mg, once per day for 90-days.

Participants will be asked to visit the laboratory (KSU Human Performance Laboratory) on 2 separate occasions for pre- and post-testing visits consisting of body composition measurements and blood draws by a CITI approved/IRB approved research team member trained in phlebotomy under the supervision of Dr. VanDusseldorp.

ELIGIBILITY:
Inclusion Criteria:

* Clinically defined as postmenopausal (absence of menstrual cycle for 12 months without contraceptives or the surgical removal of the reproductive organs)
* Activity levels ranging from sedentary to recreationally active were included in the study.

Exclusion Criteria:

* Hyper- or hypothyroidism (uncontrolled)
* Hyper- or hypoparathyroidism
* Gastrointestinal disorders
* Renal disorders
* Orthopedic disorders
* Rheumatological disorders
* Immunological disorders
* Type I diabetic
* Being treated with any diabetic injectable medication(s).
* Taking any non-steroidal, steroidal, or anti-inflammatory drugs
* Currently, or in the past 1 month, were consuming daily calcium
* Currently, or in the past 1 month, were consuming more than 5,000 IU's of vitamin D supplements
* Taking any anti-obesity medications
* Taking any osteoporotic medication(s)
* Taking any long-term antibiotics.
* Current smoker
* Diagnosed with osteoporosis, or if their BMD was equal to, or fell below -2.50 via dual x-ray absorptiometry (DXA) during visit 1
* Involved in heavy resistance training
* Began a new unaccustomed exercise routine during the 90-days
* Allergies to food(s) rich in QUE such as onions, apples, or berries; or if they were unwilling to avoid quercetin-containing foods.

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2019-08-27 (Actual); Primary Completion 2020-04-27 (Actual); Study Completion 2020-04-27 (Actual)

PRIMARY OUTCOMES:
Osteocalcin ng/mL | 90-days
  Bone formation marker
PINP ug/L | 90-days
  Procollagen type-I N-terminal propeptide. Bone formation marker.
CTX ng/L | 90-days
  Type-I collagen cross-linked C-terminal telopeptide. Bone resorption marker.
IL-6 pg/mL | 90-days
  Interleukin-6 inflammatory marker.
TNF-alpha pg/mL | 90-days
  Tumor necrosis factor-alpha inflammatory marker
CRP mg/L | 90-days
  C-reactive protein inflammatory marker.
FBG mg/dl | 90-days
  Fasting blood glucose
BMD g/cm^2 | 90-days
  Total, lumbar, right and left femur, and left forearm bone mineral density

SECONDARY OUTCOMES:
Body composition | 90-days
  body fat percentage
Timed up and go (seconds) | 90-days
  Physical function test
Dominant handgrip strength (kg) | 90-days
  Physical function test

CONTACTS AND LOCATIONS:
Locations (1):
- Kennesaw State University, Kennesaw, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bailly AR, Hester GM, Alesi MG, Buresh RJ, Feito Y, Mermier CM, Ducharme JB, VanDusseldorp TA. Quercetins efficacy on bone and inflammatory markers, body composition, and physical function in postmenopausal women. J Bone Miner Metab. 2025 May;43(3):304-314. doi: 10.1007/s00774-025-01592-0. Epub 2025 Mar 7. PMID 40053115